CLINICAL TRIAL: NCT07046013
Title: Relation Between Serum Lactate Dehydrogenase and Immune Thrombocytopenia
Brief Title: Level of Serum Lactate Dehydrogenase in Immune Thrombocytopenia
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Mahmoud Fahmy, Principal investigator, Sohag University
Other Study IDs: Soh-Med-25-5-7MS
Record Dates: First submitted 2025-06-14; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lactate dehydrogenase — It's elevation at the time of diagnosis

SUMMARY:
Assessment of relation between serum lactate dehydrogenase and immune thrombocytopenia

DETAILED DESCRIPTION:
Immune thrombocytopenia is an autoimmune disorder defined by a significantly reduced number of platelets in blood circulation.

Lactate dehydrogenase is a group of oxidoreductase isoenzymes catalyzing the reversible reaction between pyruvate and lactate.

The LDH was found to be moderately high in patients with immune thrombocytopenia at the time of diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Thrombocytopenia patients at the time of diagnosis.

Exclusion Criteria:

* bone fractures _ bone diseases_ malignancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sample collected from people newly diagnosed Immune thrombocytopenia at the time of diagnosis.
  Laboratory investigations: LDH_CBC_ESR_Bone marrow aspirate
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Relation between serum lactate dehydrogenase and immune thrombocytopenia | About 2 years

IPD SHARING:
Plan to Share IPD: Undecided